CLINICAL TRIAL: NCT01033630
Title: A Novel Randomized Double-Blind Placebo-Control Clinical Trial in High-Risk Hypertensive Subjects
Brief Title: Cardiovascular-Protective Effects of Herbal Medicine Danshen-Gegen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Prof. Thomas Yan Keung Chan, Department of Medicine and Therapeutics, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRE2005123T
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2006-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Danshen-Gegen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Image-matched placebo of active treatment
  Interventions: Drug: Placebo
- D&G 1g (Active Comparator): Randomly allocated into three groups, D&G capsule 1g/day
  Interventions: Drug: D&G 1g
- D&G 2g (Active Comparator): Randomly allocated into three groups, D&G capsule 2g/day
  Interventions: Drug: D&G 2g

INTERVENTIONS:
Drug: D&G 2g — Danshen consists of the dried root and rhizome of the perennial herb Salvia miltiorrhiza Bge. Gegen is the dried roots of Pueraria lobata (willd.). The combination in the ratio of 7:3 of the raw herbs. Capsule form, Orally taken 2g per Day
  Other Names: Danshen Gegen
  Arms: D&G 2g
Drug: D&G 1g — Danshen consists of the dried root and rhizome of the perennial herb Salvia miltiorrhiza Bge. Gegen is the dried roots of Pueraria lobata (willd.). The combination in the ratio of 7:3 of the raw herbs. Capsule form, Orally taken 1g per Day
  Other Names: Danshen Gegen
  Arms: D&G 1g
Drug: Placebo — Image-matched placebo, made with starch.
  Arms: Placebo

SUMMARY:
Atherosclerosis (in particular stroke and heart attack) is the most important health issue in modernized society and high blood pressure is an important predisposing factor. Hypertensive subjects with other chronic disease such as diabetes mellitus or impaired renal function are particularly vulnerable to these atherosclerotic complications in spite of standard antihypertensive therapies.

Danshen and Gegen are commonly used in Chinese materia medica as treatment for cardiac symptoms and atherosclerosis-related disorders.

The objective of this study is to test Danshen and Gegen as an cardiovascular-protective adjunctive regimen to prevent high-risk hypertensive cohort from primary atherosclerosis.

DETAILED DESCRIPTION:
Danshen and Gegen (D&G) are two traditional herbal medicines used for cardiac symptoms in ancient Chinese medicinal literature. Recent studies suggest their therapeutic effects in blood pressure and lipid-lowering, anti-oxidation, microcirculation-promoting, foam cells-modulation and have beneficial effects on atherogenic process in coronary patients.

To evaluate the potential of D&G in primary atherosclerosis prevention in high risk hypertension. Patients with high risk hypertension associated with left ventricular hypertrophy, diabetes mellitus and renal insufficiency were randomized to receive D&G herbal capsules (2gm/day), or (1gm/day) or identical placebo capsules in double-blind and parallel fashion for 12 months on top of their anti-hypertensive treatments. Flow-mediated dilation (endothelium-dependent dilation, FMD) and nitroglycerin-induced dilation (endothelium-independent dilation, NTG) of brachial artery, and carotid intima-media thickness (surrogate atherosclerosis marker, IMT) were measured by high resolution B-mode ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* High-risk hypertension: Asymptomatic hypertensive (pretreatment BP>160/95mmHg) subjects, currently blood pressure under control (BP<140/90mmHg),
* Aged 35-70 years
* With either (i)left ventricular hypertrophy on ECG or echocardiographic criteria, (ii) diabetes mellitus, or (iii) mild renal impairment (plasma creatinine 120-250µmol/l)

Exclusion Criteria:

* Known intolerance to D&G due to adverse effect, patients with bleeding, disorders or on long-term anticoagulation.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Ultrasound study for measuring carotid intima-media thickening (IMT) | 1 year

SECONDARY OUTCOMES:
Blood tests: lipids, creatinine, glucose, fibrinogen, hs-CRP and haemoglobin A1-C Physical examination: Blood pressure, weight, height, body mass index, hip waist ratio | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas YK Chan, Prof., Principal Investigator — Department of Medicine & Therapeutics, Prince of Wales hospital
Locations (3):
- Hong Kong (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Yan Chai Hospital, Hong Kong

REFERENCES:
- [Background] Bots ML, Hoes AW, Koudstaal PJ, Hofman A, Grobbee DE. Common carotid intima-media thickness and risk of stroke and myocardial infarction: the Rotterdam Study. Circulation. 1997 Sep 2;96(5):1432-7. doi: 10.1161/01.cir.96.5.1432. PMID 9315528
- [Background] O'Leary DH, Polak JF, Kronmal RA, Manolio TA, Burke GL, Wolfson SK Jr. Carotid-artery intima and media thickness as a risk factor for myocardial infarction and stroke in older adults. Cardiovascular Health Study Collaborative Research Group. N Engl J Med. 1999 Jan 7;340(1):14-22. doi: 10.1056/NEJM199901073400103. PMID 9878640
- [Background] Woo KS, Chook P, Raitakari OT, McQuillan B, Feng JZ, Celermajer DS. Westernization of Chinese adults and increased subclinical atherosclerosis. Arterioscler Thromb Vasc Biol. 1999 Oct;19(10):2487-93. doi: 10.1161/01.atv.19.10.2487. PMID 10521379
- [Background] Sieveking DP, Woo KS, Fung KP, Lundman P, Nakhla S, Celermajer DS. Chinese herbs Danshen and Gegen modulate key early atherogenic events in vitro. Int J Cardiol. 2005 Oct 20;105(1):40-5. doi: 10.1016/j.ijcard.2004.10.052. PMID 16207543